CLINICAL TRIAL: NCT00866645
Title: A Randomized Blind Parallel Intramuscular Haloperidol-Controlled Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Intramuscular Levosulpiride in the Treatment of Chinese Patients With Agitation Of Schizophrenia
Brief Title: A Study To Evaluate The Efficacy And Safety Of Intramuscular Levosulpiride In Patients With Agitation Of Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Hotmed Sciences Co.,LTD (Unknown)
Responsible Party: GU, Niufan, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004L03556; SMHC-100
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Agitation
Keywords: Agitation; Schizophrenia; Randomized; Blind; Parallel; Intramuscular Haloperidol; Controlled; Multicenter; Clinical Trial; Efficacy; Safety; Intramuscular Levosulpiride; Chinese; PANSS-EC; ACES; CGI; BPRS; PANSS; RSESE; BAS
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intramuscular Levosulpiride
  Interventions: Drug: Intramuscular Levosulpiride
- 2 (Active Comparator): Intramuscular Haloperidol
  Interventions: Drug: Intramuscular Haloperidol

INTERVENTIONS:
Drug: Intramuscular Haloperidol — 1ml：5mg/ampoul the recommended dose is 10 mg per day administered. Doses of 10 mg may be administered 5mg bid with an interval longer than 4 hours for 3 days.
  Other Names: Intramuscular Haloperidol parenteral solution
  Arms: 2
Drug: Intramuscular Levosulpiride — 2ml：50mg/ampoul the recommended dose is 100 mg per day administered. Doses of 100 mg may be administered 50mg bid with an interval longer than 4 hours for 3 days.
  Other Names: Intramuscular Levosulpiride parenteral solution
  Arms: 1

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of Intramuscular Levosulpiride in the treatment of Chinese patients with Agitation Of Schizophrenia compared with Intramuscular Haloperidol by evaluating the change of PANSS-EC total scores at end of study (72 hours after first dosing) from baseline.

DETAILED DESCRIPTION:
Secondary Outcome Measures:

To evaluate the change of Agitation Calmness Evaluation Scale(ACES), Clinical Global Impression(CGI, including CGI-S and CGI-I),PANSS total scores,Brief Psychiatric Rating Scale(BPRS) total scores and every item of PANSS-EC from baseline to the end of study (Time Frame: 72 hours) [ Designated as safety issue: No ]

To evaluate the change of patients' main complain, physical examination, lab and ECG tests, AE、Rating Scale for Extrapyramidal Side Effect(RSESE) and Barnes Akathisia Scale(BAS)from baseline to the end of study (Time Frame: 72 hours) [ Designated as safety issue: Yes ]

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese inpatients(are required to stay at hospital during the study) aged 18-65 years
* Patients meeting the DSM-IV criteria for schizophrenia or schizophreniform psychosis
* Agitated with a minimum total score of ≧ 15 on the five items of the PANSS-EC and at least one individual item score of ≧ 5 or two item score of ≧ 4 using the 1-7 scoring system
* ACES≤3
* Written informed consent provided by patients' legal representative

Exclusion Criteria:

* Investigator and his/her relatives
* Participation in another drug trial within 3 months prior enrolment into this study
* Female patients during their pregnant and lactation period
* Any currently severe unstable medical illness or disease would affect assessment for this study, including epilepsy, angle closure glaucoma, disease of liver, kidney, gastrointestinal tract, respiratory system, cardiovascular system(including Ischemic Heart Disease), endocrine system, nervous system, immune or hematological system etc.
* A significantly clinical abnormal value in ECG or lab results,ALT and AST values in the liver function test exceeding two times of the upper limits of normal values, urea nitrogen value arising up to 1.2 times of the upper limits of normal values, creatinine or serum potassium exceeding normal values
* With a family history of sudden death
* Meet the DSM-IV criteria for substance abuse within 1 year prior enrolment
* Regularly use antipsychotics(clozapine within 90 days), antidepressants, mood stabilizers, anti-epileptics or prolonged-action preparations within 2 weeks prior enrolment
* Use of Electroconvulsive therapy within 30 days prior enrolment
* Systematically use of sulpiride, levosulpiride or haloperidol therapy within 30 days prior enrolment
* History of or current neuroleptic malignant syndrome, severe EPS, significant tardive dyskinesia
* Severe suicide attempt
* Known hypersensitivity to sulpiride, levosulpiride or haloperidol, or history of severe drug hypersensitivity or hypersensitivity to more than 2 drugs
* Use of psychotropics(except permitted drugs) within 12 hours prior enrolment
* Known lack of efficacy to levosulpiride or haloperidol by formal treatment before
* Organic mental disorders, including Mental retardation
* History of psychosurgery treatment
* Patients can not comply with study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
the change of PANSS-EC total scores | from baseline to the end of study(72 hours after first dosing)

SECONDARY OUTCOMES:
the change of Agitation Calmness Evaluation Scale(ACES) | from baseline to the end of study (72 hours after first dosing)
The Change of Clinical Global Impression(CGI, including CGI-S and CGI-I) | from baseline to the end of study (72 hours after first dosing)
the change of PANSS total scores | from baseline to the end of study (72 hours after first dosing)
the change of Brief Psychiatric Rating Scale(BPRS) total scores | from baseline to the end of study (72 hours after first dosing)
the change of every item of PANSS-EC | from baseline to the end of study (72 hours after first dosing)
the change of Rating Scale for Extrapyramidal Side Effect(RSESE) | from baseline to the end of study (72 hours after first dosing)
the change of Barnes Akathisia Scale(BAS) | from baseline to the end of study (72 hours after first dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD,PhD, Study Director — Drug Clinical Trial Office, Shanghai Mental Health Center
Locations (5):
- China (5):
  - Hebei Mental Health Center, Baoding, Hebei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Xi'an Mental Health Center, Xi'an, Shaanxi
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - The First Affilliated Hospital Of Kunming Medical College, Kunming, Yunnan